CLINICAL TRIAL: NCT07192952
Title: A Phase 3, Single-arm, Open-label Extension Study to Evaluate the Safety of Finerenone in Addition to Standard of Care, in Pediatric Heart Failure Patients, From Birth to 18 Years of Age, With Left Ventricular Systolic Dysfunction (LVSD)
Brief Title: A Study to Learn More About How Safe Finerenone is, When it is Taken for a Longer Time With Standard Treatment, in Children and Young Adults With Heart Failure and Left Ventricular Systolic Dysfunction
Acronym: FIORELLO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21467; 2024-519830-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Left Ventricular Systolic Dysfunction; Heart Failure (Pediatric)
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Finerenone Open-Label Safety Extension (Experimental): Participants will receive finerenone treatment.
  Interventions: Drug: Finerenone (Kerendia, BAY94-8862)

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY94-8862) — Finerenone in different doses, treatment duration will be 270±7 days.

SUMMARY:
Researchers are looking for a better way to treat children and young adults who have heart failure with left ventricular systolic dysfunction (LVSD). Heart failure with left ventricular systolic dysfunction (LVSD) is a condition where the left side of the heart is weak and struggles to pump blood effectively, leading to symptoms like shortness of breath, fatigue, and poor growth.

The study treatment, finerenone (also called BAY94-8862), is under development to treat newborns, children, and young adults with heart failure and LVSD. It works by blocking a protein that contributes to inflammation, scarring, and thickening in the heart and blood vessels, which may help the heart pump more blood effectively.

The main purpose of this study is to learn about how safe finerenone is and how well it works in the long-term treatment of heart failure and LVSD.

To understand how safe the treatment is, the study team will gather information on the number of patients who experience medical problems after taking finerenone, also known as "treatment emergent adverse events" (TEAEs). Additionally, they will collect blood samples to measure levels of an electrolyte called potassium and monitor blood pressure. They will also assess kidneys function using the estimated glomerular filtration rate (eGFR).

In this study, which is an extension of the earlier done FIORE study, finerenone will also be studied in newly enrolled newborns under 6 months with heart failure and LVSD and children and young adults from the FIORE study. The participants will be aged from newborns up to 18 years. All the participants will continue to receive their standard treatment as routine care for heart failure, along with finerenone during the study.

The participants will be in the study for around 10 to 11 months, depending on whether they rolled-over from the FIORE study or are newly enrolled newborns and infants <6 months of age. They will take study treatment for up to 9 months. During this period, at least 6 visits are planned for participants. During these visits, the study team will:

* have their blood pressure, heart rate, temperature, respiratory rate, height and weight measured
* have blood samples taken
* have physical examinations
* have their heart examined by an electrocardiogram and echocardiography
* answer questions about their medication and whether they have any adverse events, or have their parents or guardians' answer
* for newborns and infants, evaluate the acceptability of the study drug formulation through parents or guardians' feedback.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

The doctors will check the participants' health a month after the participants take their last treatment.

ELIGIBILITY:
Inclusion Criteria:

* For participants rolling over from randomized controlled trial (RCT): Prior participation in the finerenone Phase 3 study FIORE (21466) and not permanently discontinued from the study intervention prior to the end of treatment (EoT) visit in FIORE.
* For newly enrolled infants <6 months of age: Left ventricular systolic dysfunction (LVSD) with left ventricular ejection fraction (LVEF) ≤ 50% at screening assessed by echocardiography.
* For newly enrolled infants <6 months of age: Elevated NT-pro BNP levels (> 500 mg/L) at screening.
* For newly enrolled infants <6 months of age: Heart failure (HF) etiologies include congenital heart defects (CHD) with biventricular physiology and systemic LV; idiopathic cardiomyopathy (CM); familial/inherited and/or genetic CM; history of myocarditis (diagnosis of an acute episode at least 3 months prior to treatment assignment); neuromuscular disorder; inborn error of metabolism; mitochondrial disorder; acquired (chemotherapy, iatrogenic, infection, rheumatic, or nutritional); ischemic (e.g., Kawasaki disease and postoperative HF); LV noncompaction.
* For newly enrolled infants <6 months of age: Receiving standard of care (SoC) treatment for heart failure according to local guidelines or investigator´s discretion (on a stable regimen for 30 days before baseline).
* Newly enrolled newborns and infants < 6 months of age must have a body weight of ≥3 kg at Visit 1.

Exclusion Criteria:

* For participants rolling over from randomized controlled trial (RCT): To roll-over to FIORELLO, all participants: Potassium (K+) >5.5 mmol/L. After unblinding:

  * For participants who received finerenone in FIORE: K+ >5.5 mmol/ L
  * For participants who received placebo in FIORE: K+ >5.0 mmol/L for children ≥2 years of age, and >5.3 mmol/L for children <2 years of age (if eGFR is <60 mL/min/1.73m² for participants <2 years of age, the serum potassium threshold of >5.0 mmol/L will be used for exclusion)
* For newly enrolled newborns and infants < 6 months of age: Potassium ≥ 5.3 mmol/l (if eGFR is <60 mL/min/1.73m², the serum potassium threshold of >5.0 mmol/L will be used for exclusion).
* For participants rolling over from RCT: Severe renal dysfunction with estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m² at FIORE EoT or Visit 1.
* For newly enrolled infants < 6 months of age: Severe renal dysfunction with eGFR < 30 ml/min/1.73m2 at screening or Visit 1.
* Treatment with a mineralocorticoid receptor antagonist, other than the study intervention, (e.g., spironolactone, eplerenone) within 30 days of Visit 1.
* Requirement of any intravenous (IV) vasoactive agents; mechanical ventilation; mechanical circulatory support; sustained or symptomatic arrhythmias not controlled by drug or device therapy within 30 days prior to study treatment.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 117 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | From the start of study intervention to last study intervention (up to 277 days) + 3 days
  TEAEs will be mapped to Medical Dictionary for Regulatory Activities (MedDRA) terms.
Change in serum potassium levels | From baseline to Day 270±7
Change in systolic blood pressure (SBP) | From baseline to Day 270±7
Change in estimated glomerular filtration rate (eGFR) | From baseline to Day 270±7

SECONDARY OUTCOMES:
Change in NT-proBNP levels | From baseline to Day 270±7
Change in left ventricular systolic function | From baseline to Day 270±7
  Change measured by echocardiogram (%) from baseline to Day 270±7
Maximum observed finerenone concentration in plasma after multiple doses (Cmax, md) | Pre-dose, post-dose (1.5-5 hours after intake of intervention), up to Day 270±7
Area under the curve for finerenone concentration in plasma after multiple doses (AUCτ,md) | Pre-dose, post-dose (1.5-5 hours after intake of intervention), up to Day 270±7
Taste and Texture Questionnaire of the pediatric formulation | On Day 30±3 and Day 270±7
  For newborns and infants <6 months of age, the taste and texture of the pediatric formulation will be evaluated using the Taste and Texture Questionnaire, completed by the caregiver, or health care professional. Results for the Taste and Texture Questionnaire from newborns and infants <6 months of age who receive the pediatric formulation will be summarized descriptively.

CONTACTS AND LOCATIONS:
Locations (132):
- United States (22):
  - Children's Hospital Colorado - Anschutz Medical Campus - Cardiology, Aurora, Colorado
  - Nemours Children's Hospital - Delaware - Cardiology, Wilmington, Delaware
  - UF Health Shands Hospital - Pediatric Cardiology, Gainesville, Florida
  - Joe Dimaggio Children's Hospital - Cardiology, Hollywood, Florida
  - Emory University Hospital - Children's Healthcare of Atlanta Cardiology - Atlanta, Atlanta, Georgia
  - Riley Hospital For Children - Cardiology, Indianapolis, Indiana
  - Boston Children's Hospital - Main Campus - Cardiology, Boston, Massachusetts
  - C.S. Mott Children's Hospital - Cardiology, Ann Arbor, Michigan
  - Children's Mercy Hospital Kansas City - Cardiology, Kansas City, Missouri
  - Washington University - St. Louis Children's Hospital - Cardiology, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai - Pediatric Cardiology, New York, New York
  - Columbia University Irving Medical Center - Pediatric Cardiology, New York, New York
  - The Children's Hospital at Montefiore - Cardiology, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center | Division of Nephrology and Hypertension, Cincinnati, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Nationwide Children's Hospital - Cardiology, Columbus, Ohio
  - Children's Hospital of Philadelphia - Cardiology, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh - Cardiology, Pittsburgh, Pennsylvania
  - MUSC Shawn Jenkins Children's Hospital - Cardiology, North Charleston, South Carolina
  - Children's Medical Center Dallas - Cardiology, Dallas, Texas
  - Texas Children's Hospital - Cardiology, Houston, Texas
  - Eccles Primary Children's Outpatient Services - Cardiology, Salt Lake City, Utah
- Argentina (10):
  - Hospital de Niños Sor María Ludovica, La Plata, Buenos Aires
  - Instituto De Investigaciones Clinicas Zarate | Zarate, Argentina, Zárate, Buenos Aires
  - Consultorios Integrados Rosario | Instituto Medico de la Fundacion de Estudios Clinicos, Rosario, Santa Fe Province
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital de Pediatría Juan P. Garrahan, Buenos Aires
  - Hospital General de Ninos Pedro de Elizalde | Nephrology Department, Buenos Aires
  - Hospital General de Ninos Ricardo Gutierrez | Pediatric Nephrology Department, Ciudad Autónoma de Buenos Aire
  - Consultorios Médicos Dr. Doreski, Ciudad Autónoma de Buenos Aire
  - Sanatorio de la Cañada, Córdoba
  - Centro Cardiovascular Salta (Torzav SRL), Salta
- Austria (2):
  - Kepler Universitätsklinikum GmbH - Klinik für Kinderkardiologie, Innsbruck, Upper Austria
  - Medizinische Universität Wien - Klinik für Kinder- und Jugendheilkunde, Abteilung für Pädiatrische Kardiologie, Vienna, Vienna
- Belgium (5):
  - UZ Leuven - Pediatric Cardiology, Leuven, Flemish Brabant
  - Cliniques Universitaires St-Luc (UCL) - Pediatric Cardiology, Brussels
  - UZ Antwerpen - Pediatric Cardiology, Edegem
  - UZ Gent - Pediatric Cardiology, Ghent
  - CHC MontLegia - Pediatric Cardiology, Liège
- Brazil (10):
  - Instituto Dante Pazzanese de Cardiologia | Divisao de Pesquisa, São Paulo, Ceará
  - InCor HCFMUSP, São Paulo, Ceará
  - Hospital de Clínicas da Universidade Federal de Uberlândia Empresa Brasileira de Serviços Hospitalares - EBSERH, Uberlandia, Espírito Santo
  - Hospital Pequeno Principe, Curitiba, Estado de Bahia
  - Hospital Infantil Sabará - Instituto PENSI - Pesquisa e Ensino em Saúde Infantil, São Paulo, Minas Gerais
  - IESG - Instituto de Ensino da Saude e Gestao, São Paulo, Rio Grande do Norte
  - Santa Casa de Misericórdia de Belo Horizonte, São Paulo, Rio Grande do Sul
  - Fundação Universidade de Caxias do Sul, Marília, São Paulo
  - Centro de Pesquisa Clinica e Populacional Hospitalize, Porto Alegre, São Paulo
  - Campinas Clinical Research Institute (IPECC) | Campinas, Brazil, São Paulo, São Paulo
- Bulgaria (4):
  - National Heart Hospital (NHH) - Dept. Pediatric Cardiology, Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment 'Sveti Georgi' EAD, Plovdiv Pediatric Clinic, Plovdiv
  - Medical Center Nora- Heart ?OOD Child Cardiology, Sofia
  - University Multiprofile Hospital for Active Treatment 'Sveta Ekaterina' EAD, Sofia, Sofia
- Canada (6):
  - Stollery Children's Hospital (SCH), Edmonton, Alberta
  - BC Children's Hospital - Children's Heart Centre, Vancouver, British Columbia
  - London Health Sciences Centre - Children's Hospital, London, Ontario
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - University of Saskatchewan, Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (2):
  - Fakultní nemocnice Brno, Detská nemocnice - Pediatrická klinika, Brno
  - Fakultní nemocnice Motol a Homolka, Pracovište MOTOL - Detské kardiocentrum 2. LF UK a FN Motol, Prague
- HUS-Yhtymä, Helsingin yliopistollinen sairaala (HUS) - Uusi lastensairaala, kardiologia, Helsinki, Finland
- Germany (3):
  - Universitaetsklinikum Giessen und Marburg GmbH - Kinderherzzentrum und Zentrum für angeborene Herzfehler, Giessen, Hesse
  - Universitätsklinikum Köln - Kinderkardiologie, Cologne
  - Universitätsklinikum Tübingen, Kinderheilkunde II - Kinderkardiologie, Pulmologie, Intensivmedizin, Tübingen
- Greece (4):
  - Onassis Cardiac Surgery Center, Department of Pediatric Cardiology and Adult Congenital Heart Disease, Kallithea, Attica
  - Athens General Children's Hospital Panagioti And Aglaia Kyriakou -2nd University Department of Pediatrics, Athens
  - Athens General Children's Hospital Panagioti And Aglaia Kyriakou, Cardiology Department, Athens
  - Nosokomeio Paidon I Agia Sofia, Cardiology Department, Athens
- Gottsegen Gyorgy Orszagos Kardiovaszkularis Intezet - Gyermeksziv Kozpont, Budapest, Hungary
- Israel (5):
  - Rambam Health Corporation, Haifa
  - Edith Wolfson Medical Center (EWMC), Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Dana-Dwek Children's Hospital, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (8):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII - Cardiologia 2 - Cardiopatie Congenite del bambino e dell'adulto, Bergamo
  - Azienda Ospedaliero-Universitaria di Bologna IRCCS Policlinico Sant'Orsola-Cardiologia pediatrica ed dell'età evolutiva, Bologna
  - IRCCS Istituto Giannina Gaslini - Cardiologia, Genova
  - ASST Grande Ospedale Metropolitano Niguarda - Struttura semplice dipartimentale cardiologia pediatrica, Milan
  - Azienda Ospedaliera Dei Colli_Monaldi - Malattie Rare e Genetiche Cardiovascolari, Naples
  - Azienda Ospedale-Università di Padova - UOC Cardiologia Pediatrica, Padua
  - Ospedale Pediatrico Bambino Gesù - Unità Terapie Cardiovascolari Avanzate, Roma
  - A.O.U. Città della Salute e della Scienza di Torino_Regina Margherita - Cadiologia pediatrica, Torino
- Mexico (8):
  - Centro de Investigación Clínica Médica y Farmacológica S.A de C.V, Guadalajara, Jalisco
  - Hospital Infantil de México "Dr. Federico Gómez", Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Pediatria, Monterrey, Nuevo León
  - Invecordis Sc., Huixquilucan, State of Mexico
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero, Tamaulipas
  - Centro de Estudios Clínicos de Querétaro S.C., Querétaro
  - Centro de Atención e Investigación Cardiovascular del Potosí S.C., San Luis Potosí City
  - Instituto Nacional de Cardiología "Ignacio Chávez", Tlalpan
- Poland (4):
  - Pomnik Centrum Zdrowia Dziecka - Klinika Kardiologii, Warsaw, Masovian Voivodeship
  - Górnoslaskie Centrum Zdrowia Dziecka im. sw. Jana Pawla II SPSK Nr 6 Slaskiego UM w Katowicach - Oddzial Kardiologii Dzieciecej, Katowice
  - Instytut Centrum Zdrowia Matki Polki w Lodzi - Klinika Kardiologii, Lódz
  - Wojewódzki Szpital Specjalistyczny we Wroclawiu Osrodek Badawczo-Rozwojowy Oddzial Kardiologii Dzieciecej, Wroclaw
- Portugal (5):
  - Department of Cardiology - Research Unit, Coimbra
  - Hospital Santa Marta | Pediatric Cardiology Department, Lisbon
  - Hospital de Santa Cruz | Pediatric Cardiology Department, Lisbon
  - Centro Materno infantil do Norte - Pediatric Cardiology, Porto
  - ULS São João - Pediatric Department, Porto
- South Korea (4):
  - Pusan National University Yangsan Children's Hospital, Yangsan, Gyeongsangnam-do
  - Seoul National University Hospital-Pediatrics Department, Jongno, Seoul
  - Severance Hospital, Yonsei University Health System-Pediatrics Department, Seodaemun
  - Samsung Medical Center-Pediatrics, Seoul
- Spain (8):
  - Hospital Sant Joan De Deu Barcelona | Cardiologia pediatrica, Esplugues de Llobregat, Barcelona
  - Hospital Universitari Vall D Hebron | Cardiologia pediatrica, Barcelona
  - Hospital Universitario Reina Sofia | Cardiologia pediatrica, Córdoba
  - Hospital Universitario Ramon Y Cajal | Cardiologia pediatrica, Madrid
  - Hospital Universitario 12 De Octubre | Cardiologia pediatrica, Madrid
  - Hospital Universitario La Paz | Cardiologia pediatrica, Madrid
  - Hospital Universitario Regional De Malaga | Cardiologia pediatrica, Málaga
  - Hospital Universitario Virgen Del Rocio S.L. | Cardiologia pediatrica, Seville
- Skånes Universitetssjukhus Lund - Barnhjärtcentrum, Lund, Skåne County, Sweden
- Taiwan (6):
  - Chang Gung Memorial Hospital (CGMH) - Kaohsiung Branch, Guishan
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Children's hospital, Taipei
- Turkey (Türkiye) (6):
  - Cukurova Universitesi Tip Fakultesi Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Bilkent Ankara
  - Marmara Uni. Tip Fak. Pendik EAH Kardiyoloji, Istanbul
  - Istanbul Mehmet Akif Ersoy Gogus Kalp Damar Cerrahisi E.A.H., Istanbul
  - Izmir Dr. Behcet Uz Cocuk Hastaliklari Hast, Izmir
- United Kingdom (7):
  - University Hospitals of Leicester NHS Trust | Leicester Children's Hospital - Children's Research Facility, Leicester, Leicestershire
  - Alder Hey Children's NHS Foundation Trust | Alder Hey Children's Hospital - Clinical Research Facility, Liverpool, Merseyside
  - Belfast Health and Social Care Trust | Royal Belfast Hospital for Sick Children - Paediatric Cardiology, Belfast, Northern Ireland
  - NHS Greater Glasgow and Clyde | Royal Hospital for Children - Glasgow Clinical Research Facility, Glasgow, Scotland
  - Newcastle upon Tyne Hospitals NHS Foundation Trust |Freeman Hospital - Children's Heart Unit, Newcastle upon Tyne, Tyne and Wear
  - Leeds Teaching Hospitals NHS Trust | Leeds Children's Hospital - Children's Research Facility, Leeds, West Yorkshire
  - University Hospitals Bristol and Weston NHS Foundation Trust | Bristol Royal Hospital for Children - Clinical Research Facility, Bristol

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.